CLINICAL TRIAL: NCT06251739
Title: Assessing Safety and Efficacy of Repurposed Oral Ivermectin in PKDL Treatment
Brief Title: Repurposing Ivermectin for PKDL Treatment
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PR-23023
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-08

CONDITIONS: Post-kala-azar Dermal Leishmaniasis
MeSH Terms: interventions — Ivermectin; miltefosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tablet Ivermectin (Active Comparator): A cumulative dose of 60 mg Oral Ivermectin monotherapy (12 mg/day) on five consecutive days (day 1 - day 5) for three consecutive months (180 mg in total)
  Interventions: Drug: Ivermectin 6 Mg Oral Tablet
- Capsule Miltefosine (Active Comparator): Oral Miltefosine monotherapy for 12 weeks. 50 mg in the morning and 50 mg in the evening with meal x 84 days (Total 100 mg/day)
  Interventions: Drug: Miltefosine Oral Capsule

INTERVENTIONS:
Drug: Ivermectin 6 Mg Oral Tablet — A cumulative dose of 60 mg Oral Ivermectin monotherapy (12 mg/day) on five consecutive days (day 1 - day 5) for three consecutive months (180 mg in total)
  Other Names: Tab. Ivera
  Arms: Tablet Ivermectin
Drug: Miltefosine Oral Capsule — Oral Miltefosine monotherapy for 12 weeks. 50 mg in the morning and 50 mg in the evening with meal x 84 days (Total 100 mg/day)
  Other Names: Cap. Miltefosine
  Arms: Capsule Miltefosine

SUMMARY:
Burden: Post-Kala-Azar Dermal Leishmaniasis (PKDL) commonly follows visceral leishmaniasis (VL) caused by Leishmania donovani. It is characterized by skin lesions in which parasites can be identified, in a patient who is otherwise fully recovered from VL or exposed to L. donovani (LD) infection. It occurs in the Indian subcontinent (mainly India and Bangladesh) as well as in Africa (mainly Sudan). It is now established that PKDL patients play an important role in transmission of LD parasite where chronic PKDL patients have been implicated in major VL outbreaks in the past. Though VL cases are in decline due to extensive programmes conducted by NKEP, PKDL cases are in the rise and VL:PKDL ratio has risen from 1:0.47 to 1:1.21 from 2016 to 2020. In this current situation, elimination of PKDL cases is of crucial importance in the current VL elimination efforts in Bangladesh as well as in the Indian subcontinent.

Knowledge gap: Currently there are no satisfactory treatments for any forms of PKDL. Both miltefosine and Ambisome® as monotherapy have shown to be effective. However, with the current recommended scheme there are some drawbacks such as the length of the treatment with miltefosine alone (8-12 weeks), toxicity related to it; a high dose Ambisome® (total dose of 20 mg/kg) given frequently in 4 divided dosage often causes adverse events (e.g. pancytopania, hypokalemia, increased creatinine level etc.). There is also the potential risk for development of resistance with miltefosine as monotherapy. Ivermectin has been proven to have a significant leishmanicidal effect by several experimental studies at higher doses without significant toxicity and may offer shorter duration of treatment thus preventing prolonged hospitalization. Another possible advantage is reduction of cost. These principles can be applied to PKDL, where the need for an ambulatory treatment with a highly safe, efficacious and user friendly regimen is even more pressing as the patients feel otherwise healthy, except for the rashes.

Relevance: This study aims primarily to improve current treatment options. In addition, this will be the first human study ever in PKDL in relation to Ivermectin, in which outcome will be described in clinical, parasitological and immunological terms. Ultimately this study findings will help National Kala-Azar Elimination Program (NKAEP) to adopt specific strategies for elimination of PKDL cases.

Hypothesis (if any): Oral ivermectin in multiple doses is safe and more effective than Miltefosine for the treatment of PKDL cases.

Objectives: To measure the safety and efficacy of Ivermectin monotherapy regimen (60 mg oral on five consecutive days, for three consecutive months) in comparison to oral Miltefosine allometric dose for twelve weeks, for treating PKDL patients in Bangladesh.

Methods: This will be a comparative, open label, non-blinded, individually randomized, proof-of-concept Clinical Trial to assess the safety and efficacy of oral Ivermectin monotherapy (5 x 12 mg daily at a total dose of 60 mg per month for three consecutive months, 180 mg in total) and Miltefosine monotherapy (50 mg twice daily for 12 weeks) in treating PKDL patients in Bangladesh. All participants will be recruited at SKKRC, Mymensingh with due consent. All patients will be followed up for 12 months. Cure assessment will be performed.

Outcome measures/variables: Safety and efficacy of Ivermectin for PKDL treatment will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed PKDL cases of either sex
* Clinically healthy except for skin lesions
* Voluntary participation through informed, voluntary written consent

Exclusion Criteria:

* Incompliance with any inclusion criteria
* Pregnant/lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-10-30 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Parasitological clearance | Within 12 months after treatment completion
  PCR in Skin samples will be negative for LD-bodies in all the Ivermectin-treated patients
Lesion Reduction | Within 12 months after treatment completion
  90 % change of PKDL lesions in patients treated with Ivermectin

SECONDARY OUTCOMES:
No Severe Adverse Events | Within 3 months following enrollment
  No Severe Adverse Events recorded in any of the patients treated with Ivermectin

OTHER OUTCOMES:
Side effects of Ivermectin | Within 3 months following enrollment
  Determine the side effects of Ivermectin when administered in multiple doses

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Mondal, MBBS,MD,PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh; Shomik Maruf, MBBS,MPH,MSc, Study Director — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Dhaka Division, Bangladesh

IPD SHARING:
Plan to Share IPD: No